CLINICAL TRIAL: NCT06331676
Title: Developing a Complex ex Vivo Endometrial Tissue Model Based on Patient Biopsies to Assess and Optimise the Response to Current and Potential Treatments for Endometriosis
Brief Title: Developing a Complex ex Vivo Endometrial Tissue Model to Improve Endometriosis Care
Acronym: OTEndo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL23_1120; 2023-A02339-36 (Other: ID RCB)
Record Dates: First submitted 2024-02-09; First posted 2024-03-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Endometriosis
Keywords: endometriosis; tissue bioengineering; hormonal therapies
MeSH Terms: conditions — Endometriosis | interventions — Tissue Banks; Data Collection

STUDY DESIGN:
Intervention Model Description: Participants enrolled in this study will be given an eutopic and ectopic endometrium biopsies, blood and peritoneal fluid sampling and should answer to a questionnaire on menstrual health and history of hormone treatments for the research purpose..
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endometriosis (Experimental): Women with endometriosis who have an indication for gynaecological surgery
  Interventions: Procedure: Tissue collection; Other: Data collection
- Control (Active Comparator): Women with no endometrial pathology who have an indication for gynaecological surgery
  Interventions: Procedure: Tissue collection; Other: Data collection

INTERVENTIONS:
Procedure: Tissue collection — Eutopic and ectopic endometrium biopsies, additional blood and peritoneal fluid sampling
Other: Data collection — Questionnaire on menstrual health and history of hormone treatments for the research purpose

SUMMARY:
Endometriosis is a chronic gynaecological disease characterised by the growth of endometrium outside the uterus. It affects 10% of childbearing age women.

There is no cure for endometriosis. Hormonal treatments should be the first line therapy. The benefit-risk ratio of symptomatic treatment with hormone therapy varies greatly from one woman to another. The pathophysiology of endometriosis and the mechanisms of action of these treatments are still poorly understood. This may be due to the lack of an optimal experimental model for studying the disease.

The aim of this project is to develop a complex ex vivo endometrial model recapitulating the organisation and properties of the human endometrium using innovative tissue bioengineering methods. This model will make it possible to develop a pre-clinical approach that predicts individual response to different types of hormonal treatment in order to optimise therapeutic choices and provide a better understanding of the effects of these treatments.

ELIGIBILITY:
Inclusion Criteria:

* Female
* People aged between 18 and 50
* Person who has or has had hormonal contraceptive treatment
* A person who has given written consent
* Person diagnosed with a benign gynaecological pathology not affecting the endometrium and requiring hysterectomy, hysteroscopy or laparoscopy or with a diagnosis of endometriosis and requiring laparoscopy or hysterectomy
* Person affiliated to the french social security

Exclusion Criteria:

* Pregnant at the time of sampling or within 3 months prior to sampling
* Breast-feeding women
* Women undergoing physiological menopause
* Anyone who has received hormonal treatment with hormones other than steroids in the three months prior to sampling
* Anyone with a non-hormonal contraceptive intrauterine device (copper coil)
* Anyone with a personal history of cancer of the breast, ovary, endometrium or cervix
* People with Lynch syndrome
* Persons under legal protection (guardianship, curatorship)
* Persons deprived of their liberty by judicial or administrative decision
* Persons with a body mass index (BMI) of less than 18.5 or more than 30

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2028-03-21 (Estimated); Study Completion 2028-03-21 (Estimated)

PRIMARY OUTCOMES:
Viability of all the cells forming the complex endometrial tissue generated ex vivo by tissue bioengineering. | through study completion, an average of 18 months
  The viability of all the cells forming the complex endometrial tissue generated ex vivo by tissue bioengineering will be assessed either by flow cytometry (labelling with propidium iodide or 7-AAD) or by immunofluorescence (with lipophilic carbocyanine dyes). The scientists involved in the project reserve the right to modify these labelling techniques and the markers mentioned, depending on the technical and logistical challenges encountered during the tissue bioengineering stages.

SECONDARY OUTCOMES:
Change in protein expression | through study completion, an average of 18 months
  Comparing changes in protein expression in the model of complex endometrial tissue generated ex vivo by tissue bioengineering (eutopic endometrium) in each donor, between control and endometriosis groups and between eutopic and ectopic endometrium in endometriosis group.
Change in gene expression | through study completion, an average of 18 months
  Comparing changes in gene expression in the model of complex endometrial tissue generated ex vivo by tissue bioengineering (eutopic endometrium) in each donor, between control and endometriosis groups and between eutopic and ectopic endometrium in endometriosis group.
Change in inflammation | through study completion, an average of 18 months
  The concentration (expressed in pg/gl) of the following cytokines will be measured using Luminex technology (Bio-Plex 200 analyser): Interleukin (IL) 1β, IL-1RA, IL-2, IL-2R, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12p40/p70, IL-13, IL-15, IL-17, Tumor Necrosis Factor TNFα, interferons (IFN) IFN-α, IFN-γ, Granulocyte-Macrophage Colony Stimulating Factor GM-CSF, Macrophage Inflammatory Protein MIP-1α, MIP-1β, Interferon gamma-induced protein 10 IP-10, Eotaxin, RANTES, and Monocyte Chemoattractant Protein-1 MCP-1.
  Changes in these inflammation markers concentration in the model of complex endometrial tissue generated ex vivo by tissue bioengineering (eutopic endometrium) in each donor, between control and endometriosis groups and between eutopic and ectopic endometrium in endometriosis group will be assessed.
Change in histological tissue structure | through study completion, an average of 18 months
  Comparing changes in histological tissue structure (density of glands open to the lumen and glands located in the basal layer of the endometrium expressed in number of glands/cm3 of tissue, measured with an haematoxiline-eosin stainings and using Image J software) in the model of complex endometrial tissue generated ex vivo by tissue bioengineering (eutopic endometrium) in each donor, between control and endometriosis groups and between eutopic and ectopic endometrium in endometriosis group.
Change in histological tissue structure | through study completion, an average of 18 months
  Comparing changes in histological tissue structure (thickness of the endometrium expressed in micrometer) in the model of complex endometrial tissue generated ex vivo by tissue bioengineering (eutopic endometrium) in each donor, between control and endometriosis groups and between eutopic and ectopic endometrium in endometriosis group.
Change in tissue elasticity | through study completion, an average of 18 months
  Comparing changes in tissue elasticity by assessing the speed of shear waves in the model of complex endometrial tissue generated ex vivo by tissue bioengineering (eutopic endometrium) in each donor, between control and endometriosis groups and between eutopic and ectopic endometrium in endometriosis group.
Change in steroid hormone physiology | At baseline
  Measurement of steroid hormones concentration levels in blood and comparison between control and endometriosis groups.
  Steroid hormones assays will be carried out using ELISA® technologies. The following hormones will be measured: prolactin, Luteinizing Hormone (LH), estradiol (E2), estrone, progesterone and Sex hormone-binding globulin SHBG. The unit of measurement is pg/ml for all hormones.
Steroid hormones in peritoneal fluid | At baseline
  Measurement of steroid hormones concentration levels in peritoneal fluid and comparison between control and endometriosis groups.
  Steroid hormones assays will be carried out using ELISA® technologies. The following hormones will be measured: prolactin, Luteinizing Hormone (LH), estradiol (E2), estrone, progesterone and Sex hormone-binding globulin SHBG. The unit of measurement is pg/ml for all hormones.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Femme Mère Enfant / GHE, Bron
  - Hôpital de la Croix-Rousse / GHN, Lyon